

Reference: PAS/L/15/0012 version 1.1

Date: 24/06/2016

# STATISTICAL ANALYSIS PLAN

Sponsor: HRA Pharma

Clinical trial protocol: 2914-012

Title: Prospective Observational Study to Assess Clinical Follow-up and Outcomes of Pregnancies Exposed to ella® (ellipse II)

Reference PAS/L/15/0012 Version 1.1

## **Sponsor**



| Company | Contact |
|--------------------------------|----------------------|
| 5 Rue Béranger,<br>75003 Paris | Christine ADELBRECHT |

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret : 432 515 914 00062 — APE : 7022 Z TVA Intracommunautaire : FR94432515914

#### **Transmitter**

| Company | Technical contact | Commercial contact | Administrative contact |
|---|---|---|---|
| SOLADIS – LYON | Ludovic BROSSAULT | François CONESA | Dominique BAUD |
| Direction des opérations | 04 72 83 86 77 | 04 72 83 86 72 | 04 72 83 86 70 |

#### **Document version**

| Version number | Date | Edition/Modification | Author |
|----------------|------------|----------------------|-------------------|
| 1.1 | 24/06/2016 | Initial Version | Ludovic BROSSAULT |

This document is confidential - Any not authorized reproduction is strictly forbidden.



Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016

Page 2 / 34

## Signature Page

| Pascale Borensztein | Date | Signature |
|---|---|---|
| Research & Development Director, HRA Pharma | 24/06/2016 | |
| Delphine Levy-Gompel | Date | Signature |
| Head of Medical Affairs, Women Health, HRA Pharma | 24 Jun 2016 | NUT |
| Christine Adelbrecht | Date | Signature / |
| Clinical Trial Coordinator, HRA Pharma | 24/06/2016 | Corningentound |
| Ludovic Brossault<br>Statistician, SOLADIS | Date 24/06/2016 | Signature |
| Pierre Clerson Clinical Study Report Medical Writer, Soladis Clinical Studies | Date 24/06/2016 | Signature |
| Babak Khoshnood | Date | Signature |
| Expert statistician, external consultant | 24/06/2016 | p. Klulus |

SARL au capital social de 50 560 € - RCS : 432 515 914 Siret : 432 515 914 00062 - APE : 7022 Z TVA Intracommunautaire : FR94432515914



## **Summary**

| 1. | INT | ROD | UCTION | 6 |
|---|---|---|---|---|
| 2. | DE | SCR | PTION OF THE STUDY | 6 |
| 2 | 2.1 | STU | DY RATIONALE | 6 |
| 2 | 2.2 | STU | DY OBJECTIVES | 7 |
| | 2.2. | .1 | PRIMARY OBJECTIVE | 7 |
| | 2.2. | .2 | SECONDARY OBJECTIVES | 7 |
| 2 | 2.3 | DES | CRIPTION OF THE OVERALL STUDY DESIGN AND PLAN | 7 |
| | 2.3 | .1 | STUDY DESIGN | 7 |
| | 2.3 | .2 | STUDY PLAN | 8 |
| 2 | 2.4 | DEF | INITION OF POPULATIONS ANALYSED | 8 |
| 3. | STI | UDY | ENDPOINTS AND ASSESSMENT METHOD | g |
| 3 | 8.1 | PRI | MARY OUTCOMES | e |
| 3 | 3.2 | SEC | ONDARY OUTCOMES | e |
| 3 | 3.3 | ENE | POINTS DERIVATION | 10 |
| | 3.3. | .1 | PRIMARY ENDPOINTS | 10 |
| | 3.3 | .2 | SECONDARY ENDPOINTS | 11 |
| | 3.3 | .3 | OTHER DEMOGRAPHIC AND CLINICAL VARIABLES | 11 |
| 4. | STI | UDY | POPULATION | 11 |
| 5. | STA | ATIS | TICAL METHODS | 12 |
| | 5.1 | | THODOLOGICAL APPROACH FOR DEMOGRAPHIC CHARACTERISTICS | |
| | 5.2 | | THODOLOGICAL APPROACH FOR PRIMARY ENDPOINTS | |
| 5 | 5.3 | | HODOLOGICAL APPROACH FOR SECONDARY ENDPOINTS | |
| | 5.4 | | NIFICANCE LEVEL | |
| 5 | 5.5 | Mıs | SING DATA | 14 |
| 5 | 5.6 | STA | TISTICAL SOFTWARE | 14 |
| 5 | 5.7 | QC | PLANS | 14 |
| 6. | RE | POR | TING CONVENTIONS | 16 |
| 6 | 6.1 | GEN | IERAL REPORTING CONVENTIONS | 16 |
| 6 | 5.2 | Ro | JNDING | 16 |
| 7. | SU | MMA | RY TABLES AND LISTINGS | 17 |
| 7 | '.1 | TAB | LES OF DEMOGRAPHIC CHARACTERISTICS | 17 |
| 7 | .2 | TAB | LES OF HISTORY OF PREGNANCY | 19 |

This document is confidential - Any not authorized reproduction is strictly forbidden.

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret : 432 515 914 00062 — APE : 7022 Z TVA Intracommunautaire : FR94432515914



## Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016

Page 4 / 34

| 7.3 | TABLES OF CHARACTERISTICS OF ELLA® INTAKE | 21 |
|---|---|---|
| 7.4 | TABLES OF CHARACTERISTICS OF PREGNANCIES | 23 |
| 7.5 | TABLE OF PATIENTS LOST TO FOLLOW-UP | 23 |
| 7.6 | RESULTS FOR PRIMARY ENDPOINTS: PREGNANCY OUTCOMES | 24 |
| 7.6 | .1 TABLE FOR THE GLOBAL POPULATION | 24 |
| 7.7 | RESULTS FOR SECONDARY ENDPOINTS | 25 |
| 7.7 | .1 Table for the overall population | 25 |
| 7.8 | RESULTS FOR CONCOMITANT MEDICATIONS | 27 |
| 7.8 | .1 TABLE FOR THE OVERALL POPULATION | 27 |
| 7.9 | Individual Listings | 28 |
| . RE | FERENCES | 34 |
| | 7.4<br>7.5<br>7.6<br>7.6<br>7.7<br>7.7<br>7.8<br>7.8<br>7.9 | 7.4 TABLES OF CHARACTERISTICS OF PREGNANCIES |

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret : 432 515 914 00062 — APE : 7022 Z TVA Intracommunautaire : FR94432515914



Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 5 / 34

## **LIST OF ABBREVIATIONS**

AE Adverse Event
BMI Body Mass Index
CI Confidence intervals

EMA European Medicine Agency
FDA Food and Drug Administration

FU Follow-Up

HCP Health Care Providers LMP Last Menstrual Period

QC Quality Control RR Risk Ratio

SAP Statistical Analysis Plan
TLF Tables, Listings and Figures

UPA Ulipristal acetate

WHO World Health Organisation

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret: 432 515 914 00062 - APE: 7022 Z

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 6 / 34

## 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the different statistical analyses which will be conducted on the study data, in conformity with the final version amended n°8.0 of the protocol 2914-012, dated the 30th March, 2015.

Any additional details or amendments will be discussed and included in a revised version of the SAP. The SAP will be finalised before database lock.

## 2. DESCRIPTION OF THE STUDY

#### 2.1 Study rationale

ella®/ellaOne® (ulipristal acetate 30 mg tablet) is a selective progesterone modulator with antagonistic and partial agonist effects at the progesterone receptor. Ulipristal acetate [17alpha-acetoxy-11beta-(4-N,N-dimethylaminophenyl)-19-norpregna-4,9-diene-3,20 dione] was initially developed at the US National Institutes of Health. The compound has been tested in an extensive battery of non-clinical and clinical studies and was approved for marketing at the dose of 30 mg (tablet) for emergency contraception up to 120 hours (5 days) under the Tradename ellaOne® in the European Union (EU/1/09/522/001) and ella® in the United States of America (NDA 022474), in May 2009 and August 2010 respectively. Initially approved as a Prescription drug, EllaOne® has been approved in Europe for marketing without prescription since January 2015.

During the evaluation process of the ella®/ellaOne® registration dossier, the EMA (European Medicines Agency) and FDA (Food and Drug Administration) requested additional information on the potential effects of ella® exposure on pregnancy course and outcome. The approval of NDA 022-474 included two post-marketing requirements (PMR 1673-1 and PMR 1673-2) as a condition of approval. PMR 1673-1 was to conduct a prospective, observational pregnancy outcome study to include fetal and neonatal outcomes and maternal pregnancy complications following a pregnancy exposed to UPA. PMR 1673-2 was to conduct a case-control study of pregnancy loss complications if a signal of concern was identified in PMR 1673-1 study. Although there were no safety signals related to pregnancy exposure to ella® from the completed phase III trials, these PMR were required by the FDA at the time of approval because there were not a sufficient number of pregnancies exposed to ella® to evaluate whether there is any fetal, neonatal or maternal risk following exposure to ella® in early pregnancy in case of emergency contraception failure or inadvertent exposure.

HRA Pharma committed to collecting information on clinical follow-up and outcomes of pregnancies that began following ella® failure as well as pregnancies inadvertently exposed to ella® by putting in place an observational study (Ellipse I), targeting 1000 investigators in Europe and the USA (Study 2914-012, Ellipse I). The main objective of the study Ellipse I was to estimate the rates of outcomes of specific events of pregnancies exposed to ella®. The secondary objectives were to collect data on birth complications of pregnancy loss in pregnancies exposed to ella® and to assess adverse events (AE) during the course of pregnancies exposed to ella®.

Recruitment of sites was very slow and difficult in the Ellipse I study and it became evident that only a limited number of pregnancies would be reported. Between 2011 and 2013; out of 219 sites initiated in Europe only 8 pregnant women were recruited. In Europe, it was decided to redirect efforts from the observational study Ellipse I towards improving the existing online European pregnancy registry. EMA thus agreed that no additional sites would be initiated and that data collection would be stopped once the improved web-based pregnancy registry would be launched.

In parallel, as per FDA requirement, decision was also taken to continue data collection in the US through the Ellipse I study and to amend the ellipse I protocol into an Ellipse II protocol (2914-012 Ellipse II) to include the web-based enrolment and prospective data collection. Pregnant Women in the US, who have been exposed to ella<sup>®</sup> during the menstrual cycle in which the pregnancy started or at any time during pregnancy will be directly enrolled in the study using a website interface that will be accessible to Health Care Professionals (HCP) and women themselves. Enrolling an exposed woman

This document is confidential - Any not authorized reproduction is strictly forbidden.



Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 7 / 34

in the study will involve completing an online questionnaire either by the HCP or directly by the woman.

In the USA, at the time of the study initiation the use of ella® was very low and limited to family planning clinics [Planned Parenthood Family planning of America (PPFA)] which typically do not follow-up women after they become pregnant. It has thus been decided to identify high-volume abortion PPFA clinics where women might have used ellaOne® to avoid a pregnancy. At these sites, such prospective studies can be performed as ultrasound reports at the time of abortion can establish living, normally-appearing pregnancies and accurate gestational age before an induced abortion taking place weeks after exposure to ellaOne®.

A total of 9 PPFA affiliates consisting of 32 abortion clinics thus accepted to participate in the Ellipse II study.

In parallel, the Ellipse II website was constantly accessible to other Health Care Professional and to any pregnant woman who has been exposed to ella<sup>®</sup> during the menstrual cycle in which the pregnancy started or at any time during pregnancy.

#### 2.2 Study objectives

#### 2.2.1 Primary objective

The primary objective of this observational study is to assess the nature and rates of pregnancy outcomes for pregnancies exposed to ella<sup>®</sup> (whether due to failure of the emergency contraception or to inadvertent exposure during pregnancy).

#### 2.2.2 Secondary objectives

The secondary objective is to assess the nature and prevalence of maternal complications in ella®-exposed pregnancies

## 2.3 Description of the overall study design and plan

#### 2.3.1 Study design

The ellipse II study is a prospective, observational study to assess clinical follow-up and outcomes of pregnancies exposed to ella<sup>®</sup>.

Enrolment will be made directly through the Website either directly by the woman or a Health Care Provider. There will be 2 different accesses: either a web-interface directly accessible by the woman for self-enrolment or an eCRF only accessible by Health Care Providers.

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret: 432 515 914 00062 - APE: 7022 Z TVA Intracommunautaire: FR94432515914

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 8 / 34

#### 2.3.2 Study plan

| | Enrolment in the study | Pregnancy<br>Course | End of pregnancy | 4 months<br>FU <sup>3</sup> |
|---|---|---|---|---|
| Written informed consent | Х | | | |
| Inclusion criteria | Х | | | |
| Pregnancy diagnosis | Χ | | | |
| ella® exposure | Χ | | | |
| Prior and concomitant medications | Х | Х | X | |
| Recreational drug use (tobacco, alcohol, illicit drugs) | Х | Х | Х | |
| Serology and prenatal tests results | Х | | | |
| Medical history | Х | | | |
| Maternal and fetal pregnancy complication | X | X | x | |
| Pregnancy outcome | | | Х | |
| Live birth follow-up | | | | Х |

## 2.4 Definition of populations analysed

Pregnancy outcomes will be described for pregnancies with known outcome (patients with missing outcomes, patients with ongoing pregnancies and patients lost to follow-up will be excluded). The proportion of patients with outcomes and lost to follow-up (or missing outcome) will be reported.



#### 3. STUDY ENDPOINTS AND ASSESSMENT METHOD

## 3.1 Primary outcomes

Outcomes to be evaluated as primary endpoints are:

- Live birth outcomes
  - Healthy baby
  - Congenital anomaly: a baby born with a congenital anomaly
  - o Neonatal death: a newborn who died during the first 28 days of life
  - Preterm birth: a baby born at less than 37 weeks of gestational age
- Pregnancy loss outcomes
  - Ectopic pregnancy: implantation of the fertilized egg and pregnancy development in a location outside the uterus and attempt to develop in this location
  - Spontaneous abortion:
    - early fetal death (i.e. < 20 completed weeks of gestation)</li>
    - missed abortion (blighted ovum)
    - not specified: all spontaneous abortions which are not early fetal death and not missed abortions
  - o Fetal death:
    - intermediate fetal death (between > 20 and <28 completed weeks of gestation)
    - late fetal death (≥ 28 completed weeks of gestation)
  - o Induced abortion can be either:
    - an induced abortion for non-medical reason
    - an induced abortion for medical reasons (termination of pregnancy for fetal anomaly, other pregnancy or maternal health complications)
  - Maternal death
- Gestational age: age of the embryo or fetus based ultrasound examination
- Normal-appearing pregnancy: medical assessment based on analysable ultrasounds results.

#### 3.2 Secondary outcomes

Outcomes to be evaluated as secondary endpoints are defined as follows:

- Maternal health complications of pregnancy are health problems of the pregnant woman that adversely affect her pregnancy, including maternal death.
- Proportion of women with ella®-exposed pregnancy complication
- Proportion of women with bleeding
- Proportion of women with infection
- Proportion of women with a need for surgical management

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret: 432 515 914 00062 - APE: 7022 Z TVA Intracommunautaire: FR94432515914

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 10 / 34

## 3.3 Endpoints derivation

## 3.3.1 Primary endpoints

The different outcomes presented above will be derived as well:

#### ✓ Live Birth outcomes

| Live births outcomes | Derivation |
|---|---|
| Proportion of live births among all pregnancy | Number of live births/total number of pregnancies |
| outcomes | |
| Proportion of healthy babies among live births | Number of healthy babies / number of live births |
| Live birth prevalence of congenital anomalies | Number of live births with congenital anomalies / |
| | number of live births |
| Live birth prevalence of other neonatal morbidity | Number of live births with neonatal morbidity |
| | (excluding congenital anomaly)/number of live |
| | births. |
| Total prevalence of congenital anomalies | Total number of congenital anomalies |
| | (terminations of pregnancy for fetal anomaly, |
| | fetal deaths, live births with congenital |
| | anomalies) / total number of births (live births + |
| | fetal deaths/stillbirths) |
| Proportion of neonatal deaths | Number of neonatal deaths / number of live births |
| Proportion of preterm births | Number of preterm births / number of live births |

#### √ Pregnancy loss outcomes

| Pregnancy loss outcomes | Derivation |
|---|---|
| Proportion of normal-appearing pregnancies (with analysable ultrasound results) before induced abortion | Number of normal-appearing pregnancies with ultrasound results compatible with normal growth and development / number of pregnancies with analysable ultrasound results which terminated by induced abortion (due to an anomaly detected, other medical reason, non-medical reason) |
| Proportion of ectopic pregnancies | Number of ectopic pregnancies / total number of pregnancies |
| Proportion of spontaneous abortions | Number of spontaneous abortions / total number of pregnancies |
| Proportion of fetal deaths | Number of fetal deaths/total number of pregnancies |
| Proportion of intermediate fetal deaths | Number of intermediate fetal deaths/total number of pregnancies |
| Proportion of late fetal deaths | Number of late fetal deaths/total number of pregnancies |
| Proportion of all induced abortions | Number of induced abortions / total number of pregnancies |
| Proportion of induced abortions for medical reason | Number of induced abortions for medical reason / total number of pregnancies |
| Proportion of induced abortion for non-medical reason | Number of induced abortions for non-medical reason / total number of pregnancies |
| Proportion of maternal deaths | Number of maternal deaths / total number of pregnancies |

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 11 / 34

#### 3.3.2 Secondary endpoints

- Proportion of women with ella®-exposed pregnancy complication = number of complications / number of pregnancies)
- Cumulative incidence of excessive bleeding episodes = number of excessive bleeding episodes / number of pregnancy losses during the study .

#### 3.3.3 Other demographic and clinical variables

Patient's age = (date of ella<sup>®</sup> intake – date of birth) / 365.25

If date of ella® intake is missing or incomplete, date of LMP will be taken into account only. If data of LMP is missing or incomplete, the date of diagnosis will be taken into account. If date of diagnosis is missing, the date of ultrasound will be taken into account. If all these dates are missing the date of pregnancy outcome (birth, induced abortion for non-medical reason, induced abortion for medical reason) or any date of examination during pregnancy (rubella test, toxoplasmosis test, prenatal test

If all these dates are missing or incomplete then age won't be recalculated and will be considered as missing.

- Time from last menstrual period (LMP) to exposure = Date of 1<sup>st</sup> ella<sup>®</sup> intake Date of first day of LMP (=date of last menstrual period)
- Exposure (repeated doses) = 1 if at least one row in the "Additional intake of ella® during pregnancy", else = 0
- BMI = weight (kg) / height (m²)

#### 4. STUDY POPULATION

The current study targets any ella<sup>®</sup>-exposed pregnant women in the US. Nevertheless, as the majority of women who become pregnant despite using an emergency contraception are attempting to avoid pregnancy, the Ellipse II study mostly targets ella<sup>®</sup>-exposed women seeking abortion services at Planned Parenthood affiliates.

The study is still ongoing until PMR fulfilment. This analysis concerns all reported pregnancies from first women included in the study through the 22<sup>nd</sup> December 2015 cut-off date and a final report will be provided at the end of study. All reported cases are included in a pooled analysis with other sources in which a single 30mg or greater doses of UPA were administered by women.

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret: 432 515 914 00062 - APE: 7022 Z TVA Intracommunautaire: FR94432515914



## 5. STATISTICAL METHODS

Given the method of patient selection for this study, the vast majority of the outcomes contained in the data base will be induced abortions for non-medical reasons. Hence, given the limited sample size for essentially all outcomes of interest, no inferential statistics will be conducted. Only descriptive statistical analyses will be performed and point estimates with 95% confidence intervals will be given for the proportions of outcomes.

Additional statistical analyses may be considered, in particular if initial results suggest that they may be feasible and necessary.

For descriptive purposes, the following statistics will be presented

**Table 5.1: Descriptive statistics summary** 

| Demographic characteristics | Categorical data | Number of subjects, number of missing data, percentage of subjects Percentages are calculated based on documented data for each outcome (non-missing observations) |
|---|---|---|
| Cital acteristics | Continuous data | Number of observations, number of missing data, mean, standard deviation, median, 1 <sup>st</sup> and third quartiles, range (minimum and maximum). |
| Primary endpoint | | Proportions (prevalence) Percentages are calculated based on documented data for each outcome |
| | Categorical data | Proportions (prevalence) Percentages are calculated based on documented data |
| Secondary endpoint | Continuous data | Number of observations, number of missing data, mean, standard deviation, median, 1 <sup>st</sup> and third quartiles, range (minimum and maximum) |

#### 5.1 Methodological approach for demographic characteristics

The following baseline characteristics data of enrolled and completed cases will be described:

- Age, as a continuous variable in years or categorical (<35 years or >=35 years groups)
- Weight in kilograms, height in meters and BMI (kg/m²)
- Sac > 20 mm (Yes, No)
- Intra-uterine pregnancy which is normal-appearing for gestational age (Yes, No, Unknown)
- Gestational age at ultrasound (weeks)
- Number of 30mg tablets of ella®
- Time from intercourse to ella® intake (hours)
- Pregnancy status before ella® intake (pregnant/not pregnant)

This document is confidential - Any not authorized reproduction is strictly forbidden.

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 13 / 34

- Pregnancy stage at ella<sup>®</sup> exposure (Before pregnancy / 1<sup>st</sup> trimester / 2<sup>nd</sup> trimester / 3<sup>rd</sup> trimester)
- How was the pregnant stage at ella® exposure determined (Ultrasound / LMP / Other)?
- time from LMP to exposure in days
- Multiple ella® intakes since LMP
- History of pregnancy (Yes, No)
- Number of previous pregnancies
- Number of live infants
- History of spontaneous abortion (miscarriage) (Yes, No)
- Number of spontaneous abortions (miscarriage)
- History of fetal death (Yes, No)
- Number of fetal deaths
- History of induced abortions for non-medical reason (Yes, No)
- Number of induced abortions for non-medical reason
- History of induced abortions for medical reason (Yes, No)
- Number of induced abortions for medical reason
- History of birth defects (Yes, No)
- Number of birth defects

Demographic characteristics of patients with known pregnancy outcome (excluding lost to follow-up patients and missing outcomes) will be described as well as those of patients where the pregnancy outcome is missing.

Patients with missing outcomes are defined as those with no pregnancy outcome ticked.

Statistical description as shown on Table 5.1 will be produced for each of these demographic characteristics.

Frequency of exposure to other drugs (other than ella®) received during pregnancy will be calculated by ATC code and drug name according to WHODRUG dictionary.

Narratives will be written for the lost follow up patients.

Moreover, baseline demographic characteristics will be presented by Pregnancy stage at ella® exposure.

In addition to these analyses, number and percent of enrolled women in each region and affiliate will be calculated on patients with known pregnancy outcome, patients with unknown pregnancy outcome and overall.

## 5.2 Methodological approach for primary endpoints

Each pregnancy outcome will be described by proportions (prevalence), as described in Table 5.1. These proportions (prevalence) of outcomes will be calculated for the overall sample.

#### 5.3 Methodological approach for secondary endpoints

The numbers of maternal and pregnancy complications will be calculated.

These analyses will be performed for the overall sample.

This document is confidential - Any not authorized reproduction is strictly forbidden.

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 14 / 34

The nature and incidence of complications of pregnancies exposed to ella® will be assessed. An individual listing will report all these individual results.

Statistical description as shown on Table 5.1 will be produced for fetal loss complications.

## 5.4 Significance level

No inferential statistical analysis will be performed.

#### 5.5 Missing data

No imputations will be performed.

#### 5.6 Statistical software

The programming of the statistical analyses will be performed by SAS® software version 9.2 or later.

## 5.7 QC plans

Two staff members are involved in the Quality Control (QC) process:

- the reviewer statistician
- the programmer

To check the quality of the analyses and programs, manual checks will be performed by reviewer.

The process for reviewer actions is the following for each Tables, Listings and Figures (TLF):

- Check of the input data base
- Manual review of SAS scripts
- · Re-run of SAS scripts
- Manual check of the SAS log
- Manual check of the SAS outputs
- Manual comparison of the SAS outputs with the TLF produced by the programmer
- QC document filling (see below)

The QC document's structure is the following:

| TLF name | Status | Comment | Correction |
|----------|--------|---------|------------|
| T001 | | | |
| T002 | | | |
| T003 | | | |
| T004 | | | |
| T005 | | | |

At the end of the process:

- If there is no issue with a TLF: Comment and Correction columns are missing and Status column is filled with "OK".
- If there is an issue with a TLF: Correction column is missing and a comment explaining the nature of the issue is written in the Comment column. Status is filled at "NOK".

The QC document will be stored on SOLADIS server. Reviewer and programmer can share this document.



Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 15 / 34

When reviewer considers it necessary to update some programs to resolve issue(s) (not necessarily after each TLF), he sends an e-mail to the programmer to adjust programs to solve the issue identified by the reviewer.

When done, the programmer filled the Correction column to "Done".

Programmer then sends an e-mail to the reviewer who re-runs the whole process for the updated TLF(s).

If the issue is solved, the reviewer fills the QC document, updating *Status*, *Comment* and *Correction* columns.

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret: 432 515 914 00062 - APE: 7022 Z

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 16 / 34

#### 6. REPORTING CONVENTIONS

## **6.1 General Reporting Conventions**

- Only standard keyboard characters should be used in tables and data listings. Special characters, such as non-printable control characters, printer specific, or font specific characters, will not be used on a table, figure, or data listing. Hexadecimal character representations are allowed (e.g., μ, α, β).
- All date values will be presented as DD/MMM/YYYY (e.g., 29/AUG/2001) format. A four-digit year is preferred for all dates.

## 6.2 Rounding

- Age as continuous variable will be truncated to become an integer variable. Example: 28.8 years
   -> 28 years.
- Integer variables (mostly duration variables) will be described with 1 decimal for mean and standard deviation estimations and no decimal for median, range and quartiles.
- Descriptive statistics for continuous variables (such as BMI) and percentages calculated for qualitative items and the various endpoints will be noted with 1 decimal.
- P-values ≥0.001 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001".</li>

SARL au capital social de 50 560 € - RCS : 432 515 914

Siret: 432 515 914 00062 - APE: 7022 Z

## 7. SUMMARY TABLES AND LISTINGS

## 7.1 Tables of demographic characteristics

Table 7.1.1: Baseline demographic – all Patients

| | Patients with known<br>pregnancy outcome<br>(TOTAL=###) | Patients with unknown pregnancy outcome (TOTAL =###) |
|---|---|---|
| Age (years) | · | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Age : n (%) | | |
| <35 years | ## (##.#) | ## (##.#) |
| >=35 years | ## (##.#) | ## (##.#) |
| Missing | ## (##.#) | ## (##.#) |
| Weight (kg) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Height (m) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| BMI (kg/m²) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##`.# ´ | ##`.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |

n: number of subjects fulfilling the item listed N: number of subjects with available data for the relevant endpoint

Table 7.2.2: Baseline demographic by pregnancy stage at ella® exposure – all Patients

| | Before pregnancy | 1st trimester (inadvertent | 2 <sup>nd</sup> trimester (inadvertent | 3 <sup>rd</sup> trimester (inadvertent | Unknown |
|---|---|---|---|---|---|
| | (treatment failure) | exposure) | exposure) | exposure) | (TOTAL=###) |
| | (TOTAL=###) | (TOTAL =###) | (TOTAL =###) | (TOTAL =###) | |
| Age (years) | | | | | |
| N | ### | ### | ### | ### | ### |
| Missing | ### | ### | ### | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) |
| Median | ##`.# | ##`.# | ##.# | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# |
| Age : n (%) | | | • | | |
| <35 years | ## (##.#) | ## (##.#) | ## (##.#) | ## (##.#) | ## (##.#) |
| >=35 years | ## (\##.# <sup>'</sup> ) | ## (\##.# <sup>'</sup> ) | ## (##.# <sup>′</sup> ) | ## (##.# <sup>°</sup> ) | ## (##.#) |
| Missing | ## (\##.# <sup>'</sup> ) | ## (\##.#) | ## (##.# <sup>′</sup> ) | ## (##.# <sup>°</sup> ) | ## (##.#) |
| Weight (kg) | , | , | , | , | ( ) |
| N V | ### | ### | ### | ### | ### |
| Missing | ### | ### | ### | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) |
| Median | ## <u>`</u> .# | ##`.# ´ | ##`.# | ## <u>`</u> # | ##`.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# |
| Height (m) | • | • | • | • | • |
| N , | ### | ### | ### | ### | ### |
| Missing | ### | ### | ### | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) |
| Median | ##`.# | ##`.# | ## <u>`</u> # | ##`.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# |
| BMI (kg/m²) | • | • | • | • | , |
| N Č | ### | ### | ### | ### | ### |
| Missing | ### | ### | ### | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# | ##`.# | ## <u>`</u> .# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# | ##.#; ##.# |

n: number of subjects fulfilling the item listed
N: number of subjects with available data for the relevant endpoint

Table 7.3.3: Baseline demographic by pregnancy stage at ella® exposure – all Patients

| | Patients with known<br>pregnancy outcome<br>(TOTAL=###) | Patients with unknown pregnancy outcome (TOTAL =###) | All patients<br>(TOTAL =###) |
|---|---|---|---|
| Region : n (%) | | | |
| Region 1 | ## (##.#) | ## (##.#) | ## (##.#) |
| Region 2 | ## (##.#) | ## (##.#) | ## (##.#) |
| <br>Missing | ## | ## | ## |
| Affiliate: n (%) | | | |
| Region 1 | ## (##.#) | ## (##.#) | ## (##.#) |
| Region 2 | ## ( <del>*</del> ##.#) | ## (##.#) | ## (##.#) |
| Missing | ## | ## | ## |

n: number of subjects fulfilling the item listed

N: number of subjects with available data for the relevant endpoint

## 7.2 Tables of history of pregnancy

Table 7.2.1. History of pregnancy – All patients

| | Patients with known<br>pregnancy outcome<br>(TOTAL=###) | Patients with unknown pregnancy outcome (TOTAL =###) |
|---|---|---|
| History of pregnancy : n (%) | · · | |
| Yes | ## (##.#) | ## (##.#) |
| No | ## (##.#) | ## (##.#) |
| Number of previous pregnancies | | |
| 1 | ## (##.#) | ## (##.#) |
| 2 | ## (##.#) | ## (##.#) |
| 3 | ## (##.#) | ## (##.#) |
| 4 | ## (##.#) | ## (##.#) |
| 5 | ## (##.#) | ## (##.#) |
| 6 | ## (##.#) | ## (##.#) |

## Table 7.2.2. History of Spontaneous abortion – All patients

Same template as Table 7.2.1

Table 7.2.3. History of Fetal death - All patients

This document is confidential - Any not authorized reproduction is strictly forbidden.

6 et 8 rue Bellecombe - 69006 LYON Tél. +33 (0) 472 838 670 - Fax : +33 (0) 472 838 671 http://www.soladis.fr - e-mail : contact@soladis.fr SARL au capital social de 50 560 € - RCS : 432 515 914

Siret : 432 515 914 00062 - APE : 7022 Z TVA Intracommunautaire : FR94432515914

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 20 / 34

Same template as Table 7.2.1

**Table 7.2.4. History of induced abortions for non-medical reason abortion – All patients** Same template as Table 7.2.1

**Table 7.2.5. History of induced abortions for medical reason – All patients** Same template as Table 7.2.1

**Table 7.2.6. History of birth defect – All patients** Same template as Table 7.2.1

SARL au capital social de 50 560 € - RCS : 432 515 914 Siret : 432 515 914 00062 - APE : 7022 Z TVA Intracommunautaire : FR94432515914

#### 7.3 Tables of characteristics of Ella® intake

Table 7.3: Ella® intake – all Patients

| | Patients with known | Patients with unknow |
|---|---|---|
| | pregnancy outcome | pregnancy outcome |
| N. J. 500 (11) ( 5 11 A | (TOTAL=###) | (TOTAL =###) |
| Number of 30mg tablets of ella® | | |
| N . | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Time from intercourse to ella® intake (in hours) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##`.# | ## <u>`</u> # |
| Min: Max | ##.#; ##.# | ##.#; ##.# |
| Time from intercourse to ella <sup>®</sup> intake (women not pregnant before ella <sup>®</sup> intake) (in hours) | · | · |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min: Max | ##.#; ##.# | ##.#; ##.# |
| Time from intercourse to ella® intake (women pregnant before ella® intake) (in | nn.n, nn.n | <i></i> , |
| hours) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min: Max | ##.#: ##.# | ##.#; ##.# |
| Pregnancy status before ella® intake : n (%) | $\pi\pi.\pi$ , $\pi\pi.\pi$ | $\pi\pi.\pi$ , $\pi\pi.\pi$ |
| | ## (##.#) | 44 (44 47) |
| Pregnant | ` , | ## (##.#) |
| Not pregnant<br>Unknown | ## (##.#) | ## (##.#)<br>## (## #\ |
| | ## (##.#) | ## (##.#) |
| Pregnancy stage at ella® exposure : n (%) | WW 700 W | "" ("" ") |
| Before pregnancy (treatment failure) | ## (##.#) | ## (##.#) |
| 1 <sup>st</sup> trimester (inadvertent exposure) | ## (##.#) | ## (##.#) |
| 2 <sup>nd</sup> trimester (inadvertent exposure) | ## (##.#) | ## (##.#) |
| 3 <sup>rd</sup> trimester (inadvertent exposure) | ## (##.#) | ## (##.#) |
| Unknown | ## (##.#) | ## (##.#) |
| How was the pregnant stage at ella® exposure determined : n (%) | | |
| Ultrasound | ## (##.#) | ## (##.#) |

This document is confidential - Any not authorized reproduction is strictly forbidden.

| LMP | ## (##.#) | ## (##.#) |
|---|---|---|
| Other | ## (##.#) | ## (##.#) |
| Time from LMP to exposure (in days) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Time from LMP to exposure (women not pregnant before ella® intake) (in days) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Time from LMP to exposure (women pregnant before ella® intake) (in days) | | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Multiple ella® intakes since her LMP : n (%) | | |
| Yes | ## (##.#) | ## (##.#) |
| No | ## (##.#) | ## (##.#) |
| Missing | ## (##.#) | ## (##.#) |

n: number of subjects fulfilling the item listed

## 7.4 Tables of characteristics of pregnancies

## Table 7.4 Characteristics of pregnancies at outcome – all patients

| | Patients with known<br>pregnancy outcome<br>(TOTAL=###) | Patients with unknown<br>pregnancy outcome<br>(TOTAL =###) |
|---|---|---|
| Gestational age at ultrasound (in weeks) | · | |
| N | ### | ### |
| Missing | ### | ### |
| Mean (SD) | ##.# (#.##) | ##.# (#.##) |
| Median | ##.# | ##.# |
| Min; Max | ##.#; ##.# | ##.#; ##.# |
| Sac > 20 mm: n (%) | | |
| Yes | ## (##.#) | ## (##.#) |
| No | ## (##.#) | ## (##.#) |
| Missing | ## (##.#) | ## (##.#) |
| Intra-uterine pregnancy which is normal-appearing for gestational age: n (%) | | |
| Yes | ## (##.#) | ## (##.#) |
| No | ## (##.#) | ## (##.#) |
| Unknown | ## (##.#) | ## (##.#) |

## 7.5 Table of patients lost to follow-up

## Table 7.5: Patients lost to follow-up – all patients

| | n/N | Proportion |
|-------------------|-------|------------|
| Lost to follow-up | xx/xx | xx.x% |

Siret: 432 515 914 00062 - APE: 7022 Z

## 7.6 Results for primary endpoints: Pregnancy outcomes

## 7.6.1 Table for the global population

Table 7.6: Primary endpoints – Patients with known pregnancy outcome

| | Primary outcome | n/N | Missing | Proportion |
|---|---|---|---|---|
| Live Birth | Proportion of live births | xx/xx | xx | xx.x% |
| | Proportion of healthy babies | xx/xx | XX | xx.x% |
| | Live births prevalence of congenital anomalies | xx/xx | xx | xx.x% |
| | Live births prevalence of other neonatal morbidity | xx/xx | xx | xx.x% |
| | Total prevalence of congenital anomalies | xx/xx | XX | xx.x% |
| | Proportion of neonatal deaths | xx/xx | XX | xx.x% |
| | Proportion of preterm births | xx/xx | XX | xx.x% |
| Pregnancy loss | Proportion of ectopic pregnancies | xx/xx | XX | xx.x% |
| | Proportion of spontaneous abortions | xx/xx | XX | xx.x% |
| | Proportion of intermediate fetal deaths | xx/xx | XX | xx.x% |
| | Proportion of late fetal deaths | xx/xx | XX | xx.x% |
| | Proportion of normal-appearing pregnancies (with analysable ultrasound results) before induced abortion | xx/xx | xx | xx.x% |
| | Proportion of all induced abortions | xx/xx | XX | xx.x% |
| | Proportion of induced abortions for non-medical reason) | xx/xx | XX | xx.x% |
| | Proportion of induced abortions for medical reason | xx/xx | XX | xx.x% |
| | Proportion of maternal deaths | xx/xx | XX | xx.x% |

## 7.7 Results for secondary endpoints

#### 7.7.1 Table for the overall population

## Table 7.7.1.1: Secondary endpoints - Healthy babies

| | Healthy babies<br>(TOTAL=###) |
|--------------------------|-------------------------------|
| Birth weight (kg) | (1011=1111) |
| N | ### |
| Missing | ### |
| Mean (SD) | ##.# (#.##) |
| Median | ##.# ´ |
| Min; Max | ##.#; ##.# |
| Delivery method : n (%) | |
| Vaginal | ## (##.#) |
| Cesarean | ## (##.#) |
| Missing | ## (##.#) |
| APGAR score at 1 minute | |
| N | ### |
| Missing | ### |
| Mean (SD) | ##.# (#.##) |
| Median | ##.# |
| Min; Max | ##.#; ##.# |
| APGAR score at 5 minutes | |
| N | ### |
| Missing | ### |
| Mean (SD) | ##.# (#.##) |
| Median | ##.# |
| Min; Max | ##.#; ##.# |

Table 7.7.1.2: Secondary endpoints - Patients with known pregnancy outcome

| Secondary<br>outcome | n/N | Missing | Proportion |
|--------------------------------------|--------|---------|------------|
| Maternal and pregnancy complications | xx/xxx | XX | xx.x% |

Table 7.7.1.3: Secondary endpoints - Fetal loss complications

| | Pregnancy los<br>(TOTAL=###) |
|---|---|
| Vaginal Bleeding : n (%) | ,, |
| Yes | ## (##.#) |
| No | ## (##.#) |
| Missing | ## (##.#) |
| Type of bleeding : n (%) | <i>"" (""")</i> |
| Spotting | ## (##.#) |
| Regular | ## (##.#) |
| Heavy | ## (##.#) |
| Missing | ## (##.#) |
| Excessive bleeding : n (%) | () |
| Yes | ## (##.#) |
| No | ## (##.#) |
| Missing | ## (##.#) |
| Duration of bleeding (days) | <i>"" (""")</i> |
| N | ### |
| Missing | ### |
| Mean (SD) | ##.# (#.##) |
| Median | ##.# |
| Min: Max | ##.#; ##.# |
| Blood transfusion performed : n (%) | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| Yes | ## (##.#) |
| No | ## (##.#) |
| Missing | ## (##.#) |
| Curettage performed : n (%) | () |
| Yes | ## (##.#) |
| No | ## (##.#) |
| Missing | ## (##.#) |
| Curettage performed : n (%) | "" (""") |
| Following the usual protocol | ## (##.#) |
| Because doctor was worried about excessive bleeding | ## (##.#) |
| Missing | ## (##.#) |
| Gestational age (weeks) | <i>"" (""")</i> |
| N | ### |
| Missing | ### |
| Mean (SD) | ##.# (#.##) |
| Median | ##.# |
| Min; Max | ##.#; ##.# |
| Infection: n (%) | $\pi\pi.\pi$ , $\pi\pi.\pi$ |
| Yes | ## (##.#) |
| No | ## (##.#) |
| Missing | ## (##.#) |
| Infection is a complication of pregnancy loss: n (%) | <del>"" ("".")</del> |

This document is confidential - Any not authorized reproduction is strictly forbidden.

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 27 / 34

| Yes | ## (##.#) |
|---------------------------|-----------|
| No | ## (##.#) |
| Unknown | ## (##.#) |
| Other complication: n (%) | |
| Yes | ## (##.#) |
| No | ## (##.#) |
| Unknown | ## (##.#) |

## 7.8 Results for concomitant medications

## 7.8.1 Table for the overall population

| Patients with at least one Conc | omitant medication | N (%) |
|---------------------------------|--------------------|-------|
| ATC code 1 | | |
| | ATC code 2 | N (%) |

SARL au capital social de 50 560 € - RCS : 432 515 914 Siret : 432 515 914 00062 - APE : 7022 Z TVA Intracommunautaire : FR94432515914

## 7.9 Individual listings

#### Listing 7.1. Listing of all pregnancies

| Subject<br>Identifier<br>for the<br>Study | Age | ВМІ | Gestational<br>age at<br>ultrasound | Date of ultrasound | Date of diagnosis | Date of<br>LMP | Expected delivery date | Number<br>of<br>tablets<br>taken | Date of<br>1st ella <sup>®</sup><br>intake | Cycle<br>day at<br>1st ella <sup>®</sup><br>intake | Date of<br>2nd<br>ella <sup>®</sup><br>intake | Cycle<br>day at<br>2 <sup>nd</sup> ella <sup>®</sup><br>intake |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

#### Listing 7.2 : Listing of patients with healthy babies

| Subject<br>Identifier<br>for the<br>Study | Age<br>calculated | Pregnant<br>at ella <sup>®</sup><br>intake | Date of conception | Pregnancy<br>term (weeks) | Number<br>of<br>babies<br>born | Baby<br>gender | Birth<br>weight<br>(kg) | Delivery<br>method | APGAR<br>score at<br>1 min | APGAR<br>score at<br>5 min |
|---|---|---|---|---|---|---|---|---|---|---|
| ID1 | XXXXX | XX | DD/MMM/YYYY | XX | XXX | Female | XX | XXXX | XX | XX |
| | | | | | | Male | XX | XXXX | XX | XX |

<sup>1</sup> baby per row

## Listing 7.3. Pregnancy information for pregnancies resulting in induced abortion for non-medical reason

| Subject<br>Identifier<br>for the<br>Study | Age<br>calculated | Gestational<br>age at<br>ultrasound | Date of<br>1st<br>ella <sup>®</sup><br>intake | Date of induced abortio n for non-medical reason | Time<br>between<br>ella <sup>®</sup><br>intake<br>and<br>outcome<br>(days) | Placenta<br>pathology<br>examination<br>performed | Examination<br>date | Examination<br>result | Pregnancy<br>term at<br>time of<br>fetal loss | Number of fetus(es) | Factors that<br>may have<br>had an<br>impact on<br>fetal loss | Other<br>comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 29 / 34

#### Listing 7.4. Induced abortions for medical reason

| Subject<br>Identifier<br>for the<br>Study | Age<br>calculated | Gestational<br>age at<br>ultrasound | Date of<br>1st<br>ella <sup>®</sup><br>intake | Date of induced abortion for medical reason | Time between ella® intake and outcome (days) | Placenta<br>pathology<br>examination<br>performed | Examination<br>date | Examination result | Pregnancy<br>term at<br>time of<br>fetal loss | Number of fetus(es) | Factors that<br>may have<br>had an<br>impact on<br>fetal loss | Other comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

#### Listing 7.5. Pregnancy information for pregnancies resulting in ectopic pregnancy

| Subject<br>Identifier<br>for the<br>Study | Age<br>calculat<br>ed | Gestati<br>onal<br>age at<br>ultrasou<br>nd | Date of<br>1st<br>ella <sup>®</sup><br>intake | Time between ella <sup>®</sup> intake and outcome (days) | Placenta<br>pathology<br>examination<br>performed | Examin<br>ation<br>date | Examinatio<br>n result | Pregnanc<br>y term at<br>time of<br>fetal loss | Number<br>of<br>fetus(es) | Factors that<br>may have had<br>an impact on<br>fetal loss | Salpingitis or<br>known tubal<br>anomaly | Previous<br>ectopic<br>pregnancy | Previous<br>tubal<br>surgery | Other<br>commen<br>ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

## Listing 7.6. Pregnancy information for pregnancies resulting in spontaneous abortion

| Subject<br>Identifier<br>for the<br>Study | Age<br>calculated | Gestational<br>age at<br>ultrasound | Date of<br>1st<br>ella <sup>®</sup><br>intake | Time between ella <sup>®</sup> intake and outcome (days) | Placenta<br>pathology<br>examination<br>performed | Examination<br>date | Examination<br>result | Pregnancy<br>term at<br>time of<br>fetal loss | Number of fetus(es) | Factors that<br>may have<br>had an<br>impact on<br>fetal loss | Other comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### Listing 7.7: Neonatal deaths - Patients with known pregnancy outcome

| ı | Subjec<br>t<br>dentifi<br>er for<br>the<br>Study | Outcom<br>e | Pregna<br>ncy<br>term | Deliv<br>ery<br>meth<br>od | Medicall<br>y<br>confirme<br>d | Age<br>calcu<br>lated | Pregnant<br>at ella <sup>®</sup><br>intake | Number<br>of<br>babies<br>born | Age of<br>neonate<br>at death<br>(days) | Cause<br>of<br>death | Relations<br>hip to<br>ella <sup>®</sup><br>intake | Autopsy<br>performed | Birth<br>weight<br>(kg) | Gender | APGAR<br>score at<br>1 min | APGAR<br>score at<br>5 min |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

<sup>1</sup> baby per row

#### Listing 7.8: Fetal loss complications - Patients with known pregnancy outcome

| Subje<br>ct<br>Identi<br>fier<br>for<br>the<br>Study | Outco<br>me | Medicall<br>y<br>confirm<br>ed | Age<br>calculat<br>ed | Pregnant<br>at ella <sup>®</sup><br>intake | Any<br>vaginal<br>bleeding? | Type of bleeding | Duration<br>of<br>bleeding | Bleedin<br>g<br>clinicall<br>y<br>excessi<br>ve | Blood<br>transfus<br>ion<br>perform<br>ed | Curetta<br>ge<br>perform<br>ed | Any<br>infectio<br>n | Locati<br>on of<br>infecti<br>on | Infecti<br>ous<br>agent | Treat<br>ment<br>given | Infecti<br>on=<br>compl<br>icatio<br>n of<br>pregn<br>ancy<br>loss | Any other complicat ion | Any other complicat ion describtio |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

## Listing 7.9. Listing of concomitant medications

| Subject<br>Identifier for<br>the Study | Pregnancy<br>outcome | Date of outcome | Date of 1st ella® intake | ATC code* | Drugname* | Indication | Intake<br>during the<br>cycle of<br>conception | Period of exposure |
|---|---|---|---|---|---|---|---|---|

<sup>\*</sup>resulting from coding with WHO Drugs dictionary

Statistical analysis plan Reference: PAS/L/15/0012 Version 1.1 of 24/06/2016 Page 31 / 34

Listing 7.10. Listing of hormonal contraception after Ella® intake in the same menstrual cycle

| Subject<br>Identifier for<br>the Study | Pregnancy outcome | Date of outcome | Date of 1st ella® intake | Medication<br>Name | Date of first<br>intake after<br>ella <sup>®</sup> intake | Route of administration |
|---|---|---|---|---|---|---|

<sup>\*</sup>resulting from coding with WHO Drugs dictionary

## Listing 7.11: Congenital anomalies - Patients with known pregnancy outcome

| Subject<br>Identifier for<br>the Study | Medically confirmed | Age calculated | Pregnant at ella <sup>®</sup> intake | Pregnancy term | Outcome | Date of conception | Date of 1st ella <sup>®</sup> intake | Date of 2nd ella <sup>®</sup> intake | Date of 3rd ella <sup>®</sup> intake |
|---|---|---|---|---|---|---|---|---|---|

| Subject<br>Identifier for<br>the Study | Age<br>calculated | Delivery<br>method | Number of babies born | List of<br>Congenital<br>anomalies | Relationship<br>to ella <sup>®</sup><br>intake | Possible cause | Gender | Birth<br>weight | APGAR<br>score at 1<br>min | APGAR<br>score at 5<br>min |
|---|---|---|---|---|---|---|---|---|---|---|

#### Listing 7.12: Maternal history - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Age<br>calculated | History of pregnancy | Number of previous pregnancies | Number<br>of live<br>infants | History of spontaneous abortion (misacarriage) | Number of spontaneous abortions | History<br>of fetal<br>death | Number<br>of fetal<br>deaths | History of induced abortions for non-medical reason | Number of induced abortions for non-medical reason |
|---|---|---|---|---|---|---|---|---|---|---|---|

| Subje<br>Identi<br>the St | fier for | History of induced abortion for medical reason | Number of induced abortions for medical reason | History of<br>birth<br>defects | Number of infants with birth defects | Specify birth defects | Description of any<br>maternal family<br>history of<br>congenital anomaly | Description of any other significant family history |
|---|---|---|---|---|---|---|---|---|

This document is confidential - Any not authorized reproduction is strictly forbidden.

### Listing 7.13: Recreational drug use - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Age<br>calculated | Drug | Y/N | Estimated weekly intake | Route of administration | 1 <sup>st</sup> trimester<br>period<br>consumption | 2 <sup>nd</sup> trimester<br>period<br>consumption | 3 <sup>rd</sup><br>trimester<br>period<br>consumption | consumption<br>throughout<br>pregnancy | Unknown<br>consumption |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ID1 | XXXXX | XX | Tobacco | X | XX | XXXX | Х | Х | Х | Х | X |
| | | | Alcohol | Χ | XX | XXXX | Х | Х | Х | Х | Х |

## Listing 7.14: Medical condition(s) during pregnancy - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Age<br>calculated | Record | Condition | Start date | Ongoing | Stop date |
|---|---|---|---|---|---|---|---|

#### Listing 7.15: Initial serology tests - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Age<br>calculated | Rubella<br>test<br>performed | Date of test | Result | Toxoplasmosis test performed | Date of test | Result |
|---|---|---|---|---|---|---|---|---|

## Listing 7.16: Prenatal tests - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Age<br>calculated | Prenatal<br>tests<br>done | Ultrasound | Ultrasound record | AFP/serum<br>markers | Amniocentesis | Reason for<br>Amniocentesis | Cordocentesis | Reason for<br>Cordocentesis | Other<br>test,<br>type | Other test, reason |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

| Subject<br>Identifier<br>for the<br>Study | Outcome | Test<br>date | Evidence of a structural defect from one or more of the prenatal tests | Specify if other | Placenta<br>pathology<br>examination<br>performed | Placenta<br>pathology<br>examination<br>Date | Placenta<br>pathology<br>examination<br>Result | Autopsy<br>performed | Autopsy<br>Date | Autopsy<br>result |
|---|---|---|---|---|---|---|---|---|---|---|

This document is confidential - Any not authorized reproduction is strictly forbidden.

Listing 7.17: Congenital anomaly detected since birth - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Number<br>of<br>babies<br>born | Baby age<br>(months) | Baby<br>height<br>(cm) | Baby<br>weight (kg) | Congenital<br>anomaly | Relationship<br>to ella <sup>®</sup><br>intake | Diagnosis<br>date | Possible causes |
|---|---|---|---|---|---|---|---|---|---|

<sup>1</sup> baby per row

Listing 7.18: Late development detected since birth - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Number<br>of<br>babies<br>born | Baby age<br>(months) | Baby<br>height<br>(cm) | Baby<br>weight (kg) | Details of<br>late<br>development<br>detected<br>since birth | Relationship<br>to ella <sup>®</sup><br>intake | Diagnosis<br>date | Possible causes |
|---|---|---|---|---|---|---|---|---|---|

<sup>1</sup> baby per row

Listing 7.19: Baby deaths - Patients with known pregnancy outcome

| Subject<br>Identifier<br>for the<br>Study | Outcome | Number<br>of<br>babies<br>born | Baby age<br>at deaths<br>(days) | Cause of death | Relationship<br>to ella <sup>®</sup><br>intake | Autopsy<br>performed | Other comments |
|---|---|---|---|---|---|---|---|





## 8. REFERENCES

[1] Newcombe R.G., Two-sided confidence intervals for the single proportion: comparison of seven methods, Statistics in Medicine, (1998) 17, 857-872